CLINICAL TRIAL: NCT04350268
Title: Exploratory Study of Wireless, Wearable Sensors at Assessing Social Interaction in Healthy Adults
Brief Title: Adult Social Interaction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: STU00209682
Record Dates: First submitted 2020-03-30; First posted 2020-04-17 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wearable sensor — Wireless sensor
  Other Names: advanced, bio-integrated wireless sensor

SUMMARY:
This study will collect vocalization data from healthy adults during regular daily activity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Subjects willing and able to comply with requirements of the protocol
* Healthy

Exclusion Criteria:

* Age <18 years old
* Subjects unwilling and able to comply with requirements of the protocol
* History of skin allergy to medical adhesive tape
* Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normal adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Speech detection | 2 years
  Talk time will be measured using computer algorithm made by the researchers in this study comparing signal to controlled, labeled signals with measured talk time.
Administration UCLA Loneliness scale. | 2 years
  Administration UCLA Loneliness scale as a proxyu assessment to measure socialization. https://fetzer.org/sites/default/files/images/stories/pdf/selfmeasures/Self_Measures_for_Loneliness_and_Interpersonal_Problems_UCLA_LONELINESS.pdf

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Evanston, Illinois, United States